CLINICAL TRIAL: NCT06112535
Title: Prospective Clinical Study to Assess the Safety and Efficacy of Versius, in Transoral Robotic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMR Surgical Ltd (Industry)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government); Sintesi Research S.r.l. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-00388
Record Dates: First submitted 2023-10-23; First posted 2023-11-01 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-03

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx; Squamous Cell Carcinoma, Unknown Primary
Keywords: TORS; robotic surgery; transoral robotic surgery
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TORS with Versius (Experimental)
  Interventions: Device: Versius Surgical System

INTERVENTIONS:
Device: Versius Surgical System — Transoral robotic surgery (TORS) using Versius Surgical System. Versius is a robot designed to help surgeons perform surgery. It consists of a set of robotic arms: one of the arms has a camera and a light source on it while the other arms each have a small surgical instrument attached at the end. The surgeon controls each of the arms with hand controllers (joysticks) and can perform surgery with them, while seeing the surgical area on a screen in front of him/her.
  The camera and instruments are inserted into the mouth and throat in order to cut out a cancerous tumour.

SUMMARY:
This is a single-arm, single site, multi-surgeon prospective feasibility study for transoral robot assisted surgery (TORS) with the Versius Surgical System. Versius is a robotic system designed to help in the accurate control of surgical instruments for minimal access ("keyhole") surgery. In TORS procedures surgical instruments are inserted through the mouth/throat to remove sick tissue rather than through skin incisions. The primary objective of this study will be to evaluate the safe use and performance of the Versius in transoral surgeries. Pre-clinical work has been conducted to ensure TORS with Versius is viable and safe; this will be one of the first in-human studies of TORS with Versius. This study will focus specifically on patients with cancerous tumours of the oropharynx (the mouth/throat) that need to be surgically removed. The safety of Versius for TORS will be mainly assessed by the rate of complications/adverse events up to 30 days after surgery, and the performance will be mainly assessed by the number of TORS cases successfully completed with Versius (i.e. without having to switch to another surgical technique).

ELIGIBILITY:
Inclusion Criteria:

1. Patient and disease factors deemed suitable for Robotic-Assisted Trans Oral Robotic Surgery (TORS) procedure using the Versius Surgical System
2. Aged 18 or over with signed, written informed consent
3. Histologically confirmed squamous cell carcinoma of the oropharynx {UICC/AJCC TNM (7) stage T1-3, N0-N2b / TNM (8) T1-3, N0-1 disease} OR Histologically confirmed squamous cell carcinoma in 1 or more cervical lymph nodes, with no discernible primary tumour (cancer unknown primary)
4. Patients considered fit for surgery and potential adjuvant treatment (WHO performance status 0-2)
5. Multidisciplinary team (MDT) decision to treat with primary surgery
6. Surgical site and anatomical factors allowing access and freedom of operating using Versius Surgical System

Exclusion Criteria:

1. T4 tumours, or T1-T3 where transoral surgery is not considered feasible due to anatomy, location, or disease factors; these may include (but not limited to) tumour visualisation, endophytic growth pattern and resulting defect functional concerns
2. Disease / anatomical factors limiting access and freedom of operating using Versius Surgical System
3. Patients with distant metastatic disease as determined by pre-operative staging
4. UICC/AJCC TNM (7) stage N2c-N3 disease; TNM (8) N2-3 disease
5. American Society of Anaesthesiologists (ASA) Class IV or above
6. WHO Performance status 3 or above
7. Unwilling or unable to sign an informed consent form
8. Morbid Obesity (BMI ≥40)
9. Active pregnancy
10. Medical Contraindication for general anaesthesia
11. Patient participation in an interventional clinical study within 30 days prior to screening, and up to 45 days post-surgery
12. Patients with a history of radiotherapy to the head or neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Incidence rate of Adverse Events | Up to 30 days post operatively
  To assess safety of TORS with Versius
Rate of successful completion of TORS without conversion | Up to completion of surgery
  To assess efficacy of TORS with Versius by the rate of successful completion of Transoral Robotic Surgery (TORS) without unplanned conversion to other transoral or open techniques

SECONDARY OUTCOMES:
Operative time | Up to completion of surgery
  Time taken to complete surgery, excluding any reconstruction
Incidence of Serious Adverse Events | Up to 30 days post operatively
  Incidence of Serious Adverse Events
Blood loss | Up to completion of surgery
  Estimated blood loss during surgery
Post-operative analgesic requirements in morphine equivalents | Up to post-surgery discharge (up to 30 days post-surgery)
  Pain medication taken post-surgery converted to morphine equivalents
Length of stay | Up to discharge (up to 30 days post-surgery)
  Length of post operative stay in hospital
Reoperation | Up to 30 days post operatively
  Emergency re-operation after initial surgery
Device deficiencies and user errors | Up to completion of surgery
  Device deficiencies and user errors
Return to oral intake | Up to post-surgery discharge (up to 30 days post-surgery)
  Amount of time after surgery before oral intake, including nasogastric tube requirement and length of use
Pathological margin | Up to 30 days post operatively
  Final pathological margin of resected specimens (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Fleming, MD PhD, Principal Investigator — ENT Department Liverpool University Hospitals NHS Foundation Trust
Locations (1):
- Liverpool Head and Neck Centre, ENT Department Liverpool University Hospitals NHS Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No